CLINICAL TRIAL: NCT05814445
Title: Comparison of Two Muscle Strengthening Programs on the Return-to-exercise Criteria in Patients With Anterior Cruciate Ligament Reconstruction
Brief Title: Muscle Strengthening and Return-to-exercise Criteria After Anterior Cruciate Ligament Reconstruction (ACLR)
Acronym: ACLR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Rehabilitacion (Other Government)
Responsible Party: Principal Investigator, Ariadna del Villar Morales, Principal Investigator, Instituto Nacional de Rehabilitacion
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27/21
Record Dates: First submitted 2023-03-30; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular exercise program (Experimental): Participants on a neuromuscular exercise program
  Interventions: Other: Neuromuscular exercise program
- Institutional exercise program (Active Comparator): Participants on an institutional exercise program
  Interventions: Other: Institutional exercise program

INTERVENTIONS:
Other: Neuromuscular exercise program — Participants will complete a neuromuscular program during 22 weeks. The program consist of isotonic open and closed kinetic chain exercises for the hip and knee, and training to improve hip and knee muscles strength, proprioception, and core stability.
  Arms: Neuromuscular exercise program
Other: Institutional exercise program — Participants will complete an institutional exercise program during 22 weeks. The program consist of isotonic open and closed kinetic chain exercises for the hip and knee, and concentric and eccentric knee exercises.
  Arms: Institutional exercise program

SUMMARY:
Anterior cruciate ligament injury is very common in recreational and elite athletes. It is considered the second most frequent pathology seeing in Sports Medicine Services. After the injury and ACLR, there is a marked decrease in the strength of the knee extensors/flexors muscles. Strength exercise programs are aimed at recovering strength and functionality, however, a low percentage of patients manage to achieve the optimal return-to-exercise criteria. Therefore, it is relevant to design and evaluate exercise programs that allow early recovery of muscle strength and knee functionality. The main purpose of this study is to investigate a neuromuscular exercise program compared with a standard institutional program in the recovery of the strength and functionality of the knee extensor/flexor muscles after ACLR.

DETAILED DESCRIPTION:
Study design: this is a 22-week, randomized trial. 62 participants will be recruited from the medical services of the National Institute of Rehabilitation (NIR).

Participants: adults between 20-40 years old, with a body mass index <30.0 kg/mˆ2, history of sports practice immediately prior to the injury, post-operated unilaterally for ACL with the hamstring autograft technique (semitendinosus-gracilis tendons), with full ranges of motion and no edema will be recruited. Participants with multi-ligament knee injuries, with more than 12 months from the injury to surgery or more than 8 months after surgery, with uncompensated metabolic diseases or acute illnesses/infections under treatment will not be recruited.

Intervention: participants will be randomized to 1) neuromuscular or 2) institutional exercise program with computer-generated random numbers. Both programs consist of isotonic open and closed kinetic chain exercises for the hip and knee. The neuromuscular program also includes exercises to improve vastus medialis and lateralis strength, hamstrings, hip flexors and extensors, proprioception, and core stability. On the other hand, the institutional program includes concentric and eccentric knee exercises. Both programs will be performed 3 days/week, 3 sets, 18-22 repetitions for each exercise; the intensity will initiate at 65-75% (1RM), and it will be increased to 75-85%; the workload will be increased 5-10% from the fifth week according to perceived exertion. The exercises will be done with both legs; however, the injured leg will be exercised complementary. The last 6 weeks of the programs correspond to functional exercises according the sport. Every training session will consist of 15 minutes of warm-up, 40-60 minutes of resistance training, and 15 minutes of cool-down; all training sessions will take place in the NIR Sports Medicine therapeutic gym.

The knee flexors/extensors muscle strength will be determined by isokinetic dynamometry (at 60°/s). The knee function will be evaluated by hop tests and agility T-test. The patient's perception of daily functional activities after ACL reconstruction will be assessed by the Lysholm knee score.

For each participant, the study length will be 22 weeks with 66 exercise sessions. The beginning of the study corresponds to session 1 of exercise. Initial evaluation will be performed 5 days prior to the start of the intervention, while final evaluations will be conducted at the end of 22 weeks of follow-up (2 days after the last day of the intervention). Data will be recorded by study investigators.

ELIGIBILITY:
Inclusion Criteria:

* History of sports practice immediately prior to the injury
* Post-operated unilaterally for ACL with the hamstring autograft technique (semitendinosus-gracilis tendons),
* Full ranges of motion and no edema
* Body mass index < 30.0 kg/mˆ2

Exclusion Criteria:

* Multi-ligament knee injuries,
* More than 12 months from the injury to surgery
* More than 8 months after surgery
* Uncompensated metabolic diseases
* Acute illnesses/infections under treatment

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Knee flexors muscle strength asymmetry | 22 weeks
  The asymmetry will be calculated as the percentage of the peak knee flexor torque in the involved limb over the peak knee flexor torque in the uninvolved limb, multiplied by 100.
  Asymmetry % = (peak flexor torque involved limb/ peak flexor torque uninvolved limb) *100
Knee extensors muscle strength asymmetry | 22 weeks
  The asymmetry will be calculated as the percentage of the peak knee extensor torque in the involved limb over the peak knee extensor torque in the uninvolved limb, multiplied by 100.
  Asymmetry % = (peak extensor torque involved limb/peak extensor torque uninvolved limb)*100
Hop distance asymmetry | 22 weeks
  The asymmetry will be calculated as the percentage of the hop distance (one leg hop, triple hop, or cross-over hop) in the involved limb over the hop distance in the uninvolved limb, multiplied by 100.
  Asymmetry % = (hop distance involved limb/hop distance uninvolved limb)*100
Agility T-test time | 22 weeks
  The time will be determined with data obtained from T-test; the fastest time will be recorded.

SECONDARY OUTCOMES:
Leg muscle quality index (MQIleg) | Baseline and 22 weeks
  The muscle quality index from legs will be calculated with data obtained by isokinetic dynamometry, and lean mass obtained by bioimpedance analysis .
  MQIleg = peak torque (Nm) / leg lean mass (kg)
Lysholm knee score | Baseline and 22 weeks
  The score consists of eighth questions rated to produce an overall score on a point scale of 0 to 100. An assignment is given as excellent for 95 to 100 points, good for 84 to 94 points, fair for 66 to 83 points, and poor for less than 65 points.

CONTACTS AND LOCATIONS:
Overall Officials: Ariadna d Morales, MD, Principal Investigator — National Institute of Rehabilitation
Locations (1):
- National Institute of Rehabilitation, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] LaBella CR, Hennrikus W, Hewett TE; Council on Sports Medicine and Fitness, and Section on Orthopaedics. Anterior cruciate ligament injuries: diagnosis, treatment, and prevention. Pediatrics. 2014 May;133(5):e1437-50. doi: 10.1542/peds.2014-0623. PMID 24777218
- [Background] van Melick N, van Cingel RE, Brooijmans F, Neeter C, van Tienen T, Hullegie W, Nijhuis-van der Sanden MW. Evidence-based clinical practice update: practice guidelines for anterior cruciate ligament rehabilitation based on a systematic review and multidisciplinary consensus. Br J Sports Med. 2016 Dec;50(24):1506-1515. doi: 10.1136/bjsports-2015-095898. Epub 2016 Aug 18. PMID 27539507
- [Background] Thomas AC, Villwock M, Wojtys EM, Palmieri-Smith RM. Lower extremity muscle strength after anterior cruciate ligament injury and reconstruction. J Athl Train. 2013 Sep-Oct;48(5):610-20. doi: 10.4085/1062-6050-48.3.23. Epub 2013 Apr 18. PMID 24067150
- [Background] Buckthorpe M, La Rosa G, Villa FD. RESTORING KNEE EXTENSOR STRENGTH AFTER ANTERIOR CRUCIATE LIGAMENT RECONSTRUCTION: A CLINICAL COMMENTARY. Int J Sports Phys Ther. 2019 Feb;14(1):159-172. PMID 30746302
- [Background] Palmieri-Smith RM, Lepley LK. Quadriceps Strength Asymmetry After Anterior Cruciate Ligament Reconstruction Alters Knee Joint Biomechanics and Functional Performance at Time of Return to Activity. Am J Sports Med. 2015 Jul;43(7):1662-9. doi: 10.1177/0363546515578252. Epub 2015 Apr 16. PMID 25883169
- [Background] Della Villa S, Boldrini L, Ricci M, Danelon F, Snyder-Mackler L, Nanni G, Roi GS. Clinical Outcomes and Return-to-Sports Participation of 50 Soccer Players After Anterior Cruciate Ligament Reconstruction Through a Sport-Specific Rehabilitation Protocol. Sports Health. 2012 Jan;4(1):17-24. doi: 10.1177/1941738111417564. PMID 23016064
- [Background] Souissi S, Wong del P, Dellal A, Croisier JL, Ellouze Z, Chamari K. Improving Functional Performance and Muscle Power 4-to-6 Months After Anterior Cruciate Ligament Reconstruction. J Sports Sci Med. 2011 Dec 1;10(4):655-64. eCollection 2011. PMID 24149555
- [Background] Cavanaugh JT, Powers M. ACL Rehabilitation Progression: Where Are We Now? Curr Rev Musculoskelet Med. 2017 Sep;10(3):289-296. doi: 10.1007/s12178-017-9426-3. PMID 28791612
- [Background] Myer GD, Brent JL, Ford KR, Hewett TE. Real-time assessment and neuromuscular training feedback techniques to prevent ACL injury in female athletes. Strength Cond J. 2011 Jun 1;33(3):21-35. doi: 10.1519/SSC.0b013e318213afa8. PMID 21643474
- [Background] Reid A, Birmingham TB, Stratford PW, Alcock GK, Giffin JR. Hop testing provides a reliable and valid outcome measure during rehabilitation after anterior cruciate ligament reconstruction. Phys Ther. 2007 Mar;87(3):337-49. doi: 10.2522/ptj.20060143. Epub 2007 Feb 20. PMID 17311886
- [Background] Noyes FR, Barber SD, Mangine RE. Abnormal lower limb symmetry determined by function hop tests after anterior cruciate ligament rupture. Am J Sports Med. 1991 Sep-Oct;19(5):513-8. doi: 10.1177/036354659101900518. PMID 1962720
- [Background] Collins NJ, Misra D, Felson DT, Crossley KM, Roos EM. Measures of knee function: International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form, Knee Injury and Osteoarthritis Outcome Score (KOOS), Knee Injury and Osteoarthritis Outcome Score Physical Function Short Form (KOOS-PS), Knee Outcome Survey Activities of Daily Living Scale (KOS-ADL), Lysholm Knee Scoring Scale, Oxford Knee Score (OKS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Activity Rating Scale (ARS), and Tegner Activity Score (TAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S208-28. doi: 10.1002/acr.20632. No abstract available. PMID 22588746
- [Background] Abrams GD, Harris JD, Gupta AK, McCormick FM, Bush-Joseph CA, Verma NN, Cole BJ, Bach BR Jr. Functional Performance Testing After Anterior Cruciate Ligament Reconstruction: A Systematic Review. Orthop J Sports Med. 2014 Jan 21;2(1):2325967113518305. doi: 10.1177/2325967113518305. eCollection 2014 Jan. PMID 26535266
- [Background] Kyritsis P, Bahr R, Landreau P, Miladi R, Witvrouw E. Likelihood of ACL graft rupture: not meeting six clinical discharge criteria before return to sport is associated with a four times greater risk of rupture. Br J Sports Med. 2016 Aug;50(15):946-51. doi: 10.1136/bjsports-2015-095908. Epub 2016 May 23. PMID 27215935
- [Background] Schmitt LC, Paterno MV, Hewett TE. The impact of quadriceps femoris strength asymmetry on functional performance at return to sport following anterior cruciate ligament reconstruction. J Orthop Sports Phys Ther. 2012 Sep;42(9):750-9. doi: 10.2519/jospt.2012.4194. Epub 2012 Jul 19. PMID 22813542
- [Background] Cristiani R, Mikkelsen C, Forssblad M, Engstrom B, Stalman A. Only one patient out of five achieves symmetrical knee function 6 months after primary anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2019 Nov;27(11):3461-3470. doi: 10.1007/s00167-019-05396-4. Epub 2019 Feb 18. PMID 30778627
- [Background] Daneshjoo A, Mokhtar A, Rahnama N, Yusof A. The effects of injury prevention warm-up programmes on knee strength in male soccer players. Biol Sport. 2013 Dec;30(4):281-8. doi: 10.5604/20831862.1077554. Epub 2013 Nov 25. PMID 24795499
- [Background] Herman K, Barton C, Malliaras P, Morrissey D. The effectiveness of neuromuscular warm-up strategies, that require no additional equipment, for preventing lower limb injuries during sports participation: a systematic review. BMC Med. 2012 Jul 19;10:75. doi: 10.1186/1741-7015-10-75. PMID 22812375
- [Background] Mandelbaum BR, Silvers HJ, Watanabe DS, Knarr JF, Thomas SD, Griffin LY, Kirkendall DT, Garrett W Jr. Effectiveness of a neuromuscular and proprioceptive training program in preventing anterior cruciate ligament injuries in female athletes: 2-year follow-up. Am J Sports Med. 2005 Jul;33(7):1003-10. doi: 10.1177/0363546504272261. Epub 2005 May 11. PMID 15888716
- [Background] Sugimoto D, Myer GD, McKeon JM, Hewett TE. Evaluation of the effectiveness of neuromuscular training to reduce anterior cruciate ligament injury in female athletes: a critical review of relative risk reduction and numbers-needed-to-treat analyses. Br J Sports Med. 2012 Nov;46(14):979-88. doi: 10.1136/bjsports-2011-090895. Epub 2012 Jun 28. PMID 22745221
- See also: Activate adult. World rugby injury prevention exercise programme. — https://australia.rugby/participate/coach/coaching-resources/world-rugby-activate